CLINICAL TRIAL: NCT06686251
Title: Evaluation of the Efficacy of Diagnostic Support Algorithms in Chest X-rays - LungAnalysis (LuAna): LuAna Stepped Wedge Trial
Brief Title: Evaluation of the Efficacy of Diagnostic Support Algorithms in Chest X-rays- LuAna Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LuAna Trial
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Consolidation; Lung Injury; Pleural Effusion; Pneumothorax; Cardiomegaly; Edema Lung
Keywords: Artificial Intelligence; Chest X-ray; Stepped wedge trial
MeSH Terms: conditions — Lung Injury; Pleural Effusion; Pneumothorax; Cardiomegaly; Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: This is a type of "stepped wedge" cluster randomized clinical trial. In the model standard of this design, interventions are implemented in the clusters randomly and graduate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App LuAna (Experimental): feedback of the artificial intelligence after the inclusion image in app LuAna.
  Interventions: Device: App LuAna

INTERVENTIONS:
Device: App LuAna — Inclusion of chest x-ray images in the LuAna app to receive feedback on lung findings.

SUMMARY:
This study aims to evaluate whether the use of AI as a physician support tool is associated with an increase in the detection rate of chest radiographic findings in adults with respiratory complaints, compared to diagnosis performed exclusively by doctors, without AI support. This is a cluster-randomized clinical trial, following the stepped wedge design, and adhering to the guidelines of the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT). In this study, the Diagnostic Support Solution for Chest X-rays - LungAnalysis (LuAna), developed by the Hospital Israelita Albert Einstein (HIAE) within the PROADI-SUS Banco de Imagens, was used.

The clinical trial will be conducted in multiple centers with a diverse population from the public health system, to ensure that the algorithms are validated across a broad demographic profile. The expected benefits are significant, providing greater security for patients, increasing doctors' confidence in interpreting chest X-rays, promoting efficiency and cost savings for healthcare services, and offering promising prospects for other AI applications in imaging diagnostics.

DETAILED DESCRIPTION:
Imaging diagnostic aid tools that use AI and facilitate the identification of findings on chest x-rays can contribute to doctors' care routines and clinicians' and radiologists' reporting routines, as these tools can allow the organization of care queues according to priorities, in addition to identifying subtle findings on the image, thereby reducing errors in reading the RXT and benefiting patients with greater agility in care and a shorter time until diagnosis. However, for reliability, these tools must undergo rigorous validation processes in large populations before implementation.

ELIGIBILITY:
Inclusion Criteria:

* Non-reported chest X-rays (XRts) of individuals aged over 18 years.
* Individuals images with respiratory complaints.
* Chest X-rays taken during the presence of these respiratory symptoms or while being followed up for respiratory disease.
* Chest X-rays taken on any X-ray machine.
* Chest X-rays that include at least one frontal view of the chest.

Exclusion Criteria:

* Those whose chest X-ray was performed due to a history of trauma, pre-operative risk assessment, lung cancer screening, or exclusively for verifying the correct positioning of a peripheral intravenous catheter (PICC).
* Chest X-rays with technical quality below the minimum required for proper interpretation and diagnosis.
* Cases without at least one frontal view.
* X-rays printed on regular paper.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1470 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate | through study completion, an average of 1 year
  Detection rate of "Radiological Findings", before and after Artificial Intelligence assistance, compared to gold standard (report validated twice by thoracic radiologists blind to the interpretation of the examining physician and AI result).

CONTACTS AND LOCATIONS:
Overall Officials: Joselisa Paiva, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- FEAS Curitiba, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No